CLINICAL TRIAL: NCT04971837
Title: Interaction Between Cannabidiol, Meal Ingestion, and Liver Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Christopher Bell, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-10634H
Record Dates: First submitted 2021-06-04; First posted 2021-07-22 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Metabolism; Liver Function; Pharmacokinetics
MeSH Terms: interventions — Cannabidiol; Gum Arabic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The CBD and placebo formulations are prepared, bottled and coded by Caliper Foods. The participants will receive a coded bottle to consume of the different formulations of CBD and placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Two Visits Including A Test Meal (Experimental): Separated by a minimum of 4 days.
  Interventions: Dietary Supplement: Cannabidiol (CBD) powder formulation; Dietary Supplement: CBD matching Placebo
- Five Visits Not Involving A Test Meal (Experimental): Separated by a minimum of 14 days.
  Interventions: Dietary Supplement: Cannabidiol (CBD) powder formulation; Dietary Supplement: Cannabidiol (CBD) Oil based tincture formulation; Dietary Supplement: Cannabidiol (CBD) Gum Arabic, maltodextrin base formulation; Dietary Supplement: Cannabidiol (CBD) Gum Arabic, sorbitol base formulation; Dietary Supplement: Cannabidiol (CBD) Isolate in water formulation

INTERVENTIONS:
Dietary Supplement: Cannabidiol (CBD) powder formulation — T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate (Formulation 725: Water soluble.Contains sorbitol)
Dietary Supplement: Cannabidiol (CBD) Oil based tincture formulation — 30 mg CBD isolate in MCT oil,1:1 ratio of CBD to Medium Chain Triglycerides oil. (Formulation 088: Not water soluble. Contains medium chain triglyceride coconut oil.)
  Arms: Five Visits Not Involving A Test Meal
Dietary Supplement: Cannabidiol (CBD) Gum Arabic, maltodextrin base formulation — 10% CBD Gum Arabic, maltodextrin base(Formulation 126: Water soluble. Contains gum arabic and maltodextrin)
  Arms: Five Visits Not Involving A Test Meal
Dietary Supplement: Cannabidiol (CBD) Gum Arabic, sorbitol base formulation — 10% CBD Gum Arabic, sorbitol base (Formulation 213: Water soluble. Contains gum arabic and sorbitol)
  Arms: Five Visits Not Involving A Test Meal
Dietary Supplement: Cannabidiol (CBD) Isolate in water formulation — Pure CBD as crystalline powder (>99% purity) (Formulation 625 Not water soluble)
  Arms: Five Visits Not Involving A Test Meal
Dietary Supplement: CBD matching Placebo — Matching Placebo
  Arms: Two Visits Including A Test Meal

SUMMARY:
According to a recent consumer poll, over 20 million Americans regularly use cannabidiol (CBD). Moreover, 64 million Americans (over 25% of the population) report trying CBD at least once within the previous 2 years. Since the passing of the 2018 Agriculture Improvement Act, the use of hemp-derived products, such as CBD, is highly prevalent across North America. The acceleration of the use of CBD has outpaced our understanding of the associated potential risks and benefits, and the way it is processed within the body.

In the current proposed project, investigators wish to continue our ongoing collaboration with Caliper Foods, a Colorado-based manufacturer of CBD products. The focus of this project is three-fold: (1) investigators will compare the pharmacokinetics of different formulations of ingestible CBD; (2) investigators will examine the potential two-way interaction between a meal and one formulation of ingestible CBD; and, (3) investigators will examine the influence of different formulations of CBD on markers of liver function.

DETAILED DESCRIPTION:
Pharmacokinetics describes the speed in which something that is ingested is made available within the body (i.e. bioavailability).There are many different preparations/formulations of CBD and they may differ from one another with regards to their pharmacokinetics. One important consideration when evaluating CBD formulations is the pharmacokinetic goal and intended use. For example, if the indication for the CBD is to treat acute pain, then a faster time to peak concentration (Tmax) and higher maximal concentration (Cmax) may be desirable, and also may help to decrease the risk of overdose due to premature repeat self administration. Alternatively, as a chronic treatment for anxiety, a larger area under the curve (AUC) may be preferable if a user follows a regular dosing schedule.

One purpose of the proposed project is to compare the pharmacokinetics of different formulations of CBD. The formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble).

Several previous studies have demonstrated an influence of eating on the pharmacokinetics of ingested CBD. The general consensus appears to be that prior ingestion of a high-fat meal increases the maximal concentration of circulating CBD (Cmax) and lowers the time to attain peak circulating concentration (Tmax).

One purpose of the proposed project is to study the influence of a standardized meal on the pharmacokinetics of a CBD formulation.

Little is known about the influence of ingested CBD on postprandial metabolism. The thermic effect of feeding (i.e. the increase in metabolic rate above resting metabolism) is considered an important physiological determinant of energy balance, and therefore also of weight gain or loss. Further, the dynamics of circulating glucose and triglycerides following a meal are reflective of metabolic health and predictive of future cardiometabolic disease risk. CBD has been purported to have a variety of beneficial physiological properties, including anti-inflammatory and antioxidant actions. Either of these individual properties alone could favorably modify postprandial metabolism, given that CBD potentially does both, it appears likely that CBD might improve the physiological regulation of postprandial metabolism.

One purpose of the proposed project is to determine the influence of CBD on postprandial metabolism.

The liver plays a critical regulatory role in postprandial metabolism, and also with the physiological processing of cannabinoids. The relationship between the use of cannabinoids and liver health is unclear. While early studies implied that exposure of the liver to very high daily dosing of cannabinoids may be detrimental, more recent studies are suggesting that some cannabinoids, including CBD, may have therapeutic potential for the treatment of non-alcoholic fatty liver disease. The acute effects of low dose CBD (e.g. 30 mg) on liver function in healthy adults have not been well described, and may be influenced by the formulation of the CBD product (i.e. whether it is water or lipid soluble).

One purpose of the proposed project is to determine the acute influence of different formulations of CBD on circulating markers of liver function.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be greater than 18 years of age
* Weigh more than 110 pounds
* Have a body mass index greater than 25kg/m^2
* Be free of any gastrointestinal or metabolic diseases
* Be able to refrain from use of any Cannabis or cannabis containing products for three days prior to participating in the study.

Exclusion Criteria:

* Less than 18 years of age
* Pregnant or breastfeeding
* Food allergies
* Autoimmune disorders or with compromised immune function,
* Celiac disease
* Inflammatory bowel Diseases
* Gastrointestinal cancers
* Diabetes
* HIV
* Adverse reactions to ingesting Cannabis spp. or cannabis-containing products (including, but not limited to, marijuana, CBD oils, or CBD/THC containing food products)
* Taking any of the follow medications: steroids, HMG-CoA reductase inhibitors, calcium channel blockers, antihistamines, HIV antivirals, immune modulators, benzodiazepines, antiarrythmics, antibiotics, anesthetics, antipsychotics, antidepressants, anti-epileptics, beta blockers, proton pump inhibitors, NSAIDs, angiotension II blockers, oral hypoglycemic agents, and sulfonylureas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2021-12-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Dept. of Health and Exercise Science, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbotts KSS, Ewell TR, Butterklee HM, Bomar MC, Akagi N, Dooley GP, Bell C. Cannabidiol and Cannabidiol Metabolites: Pharmacokinetics, Interaction with Food, and Influence on Liver Function. Nutrients. 2022 May 21;14(10):2152. doi: 10.3390/nu14102152. PMID 35631293

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Experimental: Two Visits Including A Test Meal Separated by a minimum of 4 days. Dietary Supplement: Cannabidiol (CBD) powder formulation T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate (Formulation 725: Water soluble.Contains sorbitol) Dietary Supplement: CBD matching Placebo Matching Placebo
  Experimental: Five Visits Not Involving A Test Meal Separated by a minimum of 14 days. Dietary Supplement: Cannabidiol (CBD) powder formulation T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate (Formulation 725: Water soluble.Contains sorbitol)
  Dietary Supplement: Cannabidiol (CBD) Oil based tincture formulation 30 mg CBD isolate in MCT oil,1:1 ratio of CBD to Medium Chain Triglycerides oil. (Formulation 088: Not water soluble. Contains medium chain triglyceride coconut oil.)
  Dietary Supplement: Cannabidiol (CBD) Gum Arabic, maltodextrin base formulation 10% CBD Gum Arabic, maltodextrin base(Formulation 126: Water soluble. Contains gum arabic and maltodextrin)
  Dietary Supplement: Cannabidiol (CBD) Gum Arabic, sorbitol base formulation10% CBD Gum Arabic, sorbitol base (Formulation 213: Water soluble. Contains gum arabic and sorbitol)
  Dietary Supplement: Cannabidiol (CBD) Isolate in water formulation Pure CBD as crystalline powder (>99% purity) (Formulation 625 Not water soluble)
Period: Overall Study
Arm/Group | All Study Participants
Started | 26
Formulation 126 Without Meal, | 15
Formulation 213 Without Meal | 14
Formulation 625 Without Meal | 16
Formulation 725 Without Meal | 14
Formulation 088 Without Meal, | 15
Formulation 725 With Meal | 14
Placebo With Meal | 14
Completed | 14
Not Completed | 12
Not completed — Long Term Illness | 1
Not completed — BMI too low | 9
Not completed — geographic location | 1
Not completed — Discontinued scheduling conflict | 1

BASELINE CHARACTERISTICS:
Groups:
- Over Number of Study Participants: Randomized Cross over study
Arm/Group | Over Number of Study Participants
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Time to Maximum Concentration- (Tmax) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate Tmax (minutes).
Time Frame: Venous blood will be sampled at standardized intervals: 0, 10, 20, 30, 45, 60, 120, 180, and 240 minutes and will be analyzed to compare circulating CBD concentration.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Formulation 088: Not water soluble. Contains medium chain triglyceride coconut oil.
- Formulation 126: Water soluble. Contains gum arabic and maltodextrin
- Formulation 213: Water soluble. Contains gum arabic and sorbitol
- Formulation 625: Not water soluble. Pure CBD as crystalline powder (>99% purity)
- Formulation 725: Water soluble. Contains sorbitol
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 12 | 14 | 14 | 11 | 14
minutes | 116.3 (76) | 35.4 (13.5) | 51.8 (24.2) | 129.5 (89.6) | 38.2 (24.9)

2. Primary Outcome: Pharmacokinetic Maximum Concentration-(Cmax) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate Cmax (ng/mL).
Time Frame: venous blood will be sampled at standardized intervals over 4-hours: 0, 10, 20, 30, 45, 60, 120, 180, and 240 minutes and will be analyzed to compare circulating CBD concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 12 | 14 | 14 | 11 | 14
ng/mL | 0.5 (0.2) | 3.1 (2.1) | 2.2 (2.0) | 0.4 (0.6) | 1.8 (1.5)

3. Primary Outcome: Pharmacokinetic Area Under the Curve Representing Total Cannabidiol Exposure Between 0 and 4 h (AUC 0-4) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate AUC 0-4 (min x ng/mL).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes x ng/mL
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 12 | 14 | 14 | 11 | 14
minutes x ng/mL | 62.8 (29.7) | 272.3 (176) | 208.6 (151.1) | 46 (59.4) | 177.3 (104.8)

4. Primary Outcome: Pharmacokinetic Area Under the Curve an Estimate of Total Exposure to CBD Over Time (AUC 0-inf) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate AUC 0-inf (mins x ng/mL).
Time Frame: as for outcome 2
Population: Data not collected or analyzed in groups listing 0 for overall number of participants analyzed.
Measure: Mean (Standard Deviation); unit: minutes x ng/mL
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 0 | 6 | 5 | 0 | 2
minutes x ng/mL |  | 385.2 (226.6) | 367.6 (217.1) |  | 301.6 (221.9)

5. Primary Outcome: Pharmacokinetic Amount of Time it Takes to Decrease the Circulating Concentration to Half of Its Initial Value (t1/2) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate t1/2 (mins).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 5 | 14 | 11 | 3 | 13
minutes | 280.7 (141.5) | 171.0 (129.2) | 140.5 (96.6) | 442.7 (451.0) | 133.1 (26.7)

6. Primary Outcome: Pharmacokinetic Rate at Which CBD is Absorbed Into the Body (Ka) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate Ka(1/h).
Time Frame: as for outcome 2
Population: Outcome measure not collected
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Pharmacokinetic Rate at Which CBD is Removed From the Body (Ke) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate Ke (1/h).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/h
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 5 | 14 | 11 | 3 | 13
1/h | 00.003 (.001) | .006 (.003) | .006 (.002) | 0.003 (.002) | 0.005 (.001)

8. Primary Outcome: CBD Pharmacokinetic Volume of Distribution- (Vd) for Different Formulations of CBD
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be sampled at standardized intervals over 4-hours to calculate Vd (L).
Time Frame: as for outcome 2
Population: Data not collected or analyzed in groups listing 0 for overall number of participants analyzed.
Measure: Mean (Standard Error); unit: mL, 1 L is equal to 1,000 mL
Arm/Group | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 0 | 6 | 5 | 0 | 2
mL, 1 L is equal to 1,000 mL |  | 11836405 (7642484) | 13130100 (6339554) |  | 22687960 (16435999)

9. Primary Outcome: Pharmacokinetic Parameter Tmax of a Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts the time to attain peak circulating concentration Tmax (mins).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Formulation 725
Number analyzed (Participants) | 14
minutes | 113.6 (70.5)

10. Primary Outcome: Pharmacokinetic Parameter Cmax of a Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD Cmax (ng/L).
Time Frame: venous blood will be sampled at standardized intervals over: 0, 10, 20, 30, 45, 60, 120, 180, and 240 minutes and will be analyzed to compare circulating CBD concentration.
Measure: Mean (Standard Deviation); unit: ng/mL. 1 L is equal to 1,000 mL.
Arm/Group | Formulation 725
Number analyzed (Participants) | 14
ng/mL. 1 L is equal to 1,000 mL. | 2.9 (1.3)

11. Primary Outcome: Pharmacokinetic Parameter AUC 0-4 of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD AUC 0-4 (min x ng/mL).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: min x ng/mL
Arm/Group | Formulation 725
Number analyzed (Participants) | 14
min x ng/mL | 397 (167)

12. Primary Outcome: Pharmacokinetic Parameter AUC 0-inf of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD AUC 0-inf (min x ng/mL).
Time Frame: venous blood will be sampled at standardized intervals 0, 10, 20, 30, 45, 60, 120, 180, and 240 minutes and will be analyzed to compare circulating CBD concentration.
Population: Data not Collected
Arm/Group | Formulation 725
Number analyzed (Participants) | 0

13. Primary Outcome: Pharmacokinetic Parameter t1/2 of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD t1/2 (h).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes, 1 hour is equal to 60 minutes.
Arm/Group | Formulation 725
Number analyzed (Participants) | 7
minutes, 1 hour is equal to 60 minutes. | 248.6 (304.6)

14. Primary Outcome: Pharmacokinetic Parameter Ka of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD Ka (1/h).
Time Frame: as for outcome 2
Population: Data not collected
Arm/Group | Formulation 725
Number analyzed (Participants) | 0

15. Primary Outcome: Pharmacokinetic Parameter Ke of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD Ke (1/h).
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Formulation 725
Number analyzed (Participants) | 7
1/hour | 0.005 (0.002)

16. Primary Outcome: Pharmacokinetic Parameter Vd of Formulation 725 After a Standardized Meal
Description: At the 2 randomized visits Including a Test Meal, determine if a high-fat meal impacts maximal concentration of circulating CBD Vd (L).
Time Frame: as for outcome 2
Population: Data Not Collected
Groups:
- Dietary Supplement: Cannabidiol (CBD) Isolate in Water Formulation: Formulation contains sorbitol
Arm/Group | Dietary Supplement: Cannabidiol (CBD) Isolate in Water Formulation
Number analyzed (Participants) | 0

17. Primary Outcome: Ingested CBD on Postprandial Metabolism Via Indirect Calorimetry
Description: At the 2 randomized visits Including a Test Meal Thermic Effect of Feeding (TEF) Under the Curve was calculated from standardized intervals prior to and after ingestion of a liquid meal and a single dose of Formulation 725.
Time Frame: Randomized visit Including a test meal collected during 235 minutes of TEF
Population: The thermic effect of feeding refers to the increase in energy expenditure after eating. On the X-axis, the independent variable is time, and the unit is minutes (min). On the Y-axis, the dependent variable is energy expenditure, and the unit is kilocalories per minute (kcal/min). Thus, the unit for area under the curve is kcal/min X min.
Measure: Mean (Standard Deviation); unit: (kcal/min) x min
Groups:
- Placebo: CBD-free placebo.
Arm/Group | Formulation 725 | Placebo
Number analyzed (Participants) | 14 | 14
(kcal/min) x min | 58.83 (14.3) | 55.28 (27.62)

18. Primary Outcome: Ingested CBD on Postprandial Metabolism Via Measurements of Glucose
Description: At the 2 randomized visits Including a Test Meal, glucose Area Under the Curve was calculated from standardized intervals after ingestion of a liquid meal and a single dose of Formulation 725.
Time Frame: Compare 2 randomized visits Including a test meal collected at baseline,10,20,30,45,60,90,120,150,180,210, and 240 minutes.
Measure: Mean (Standard Deviation); unit: min x mg/dL
Arm/Group | Formulation 725 | Placebo
Number analyzed (Participants) | 13 | 14
min x mg/dL | 18634.8 (2651.8) | 19001.72 (4037.1)

19. Primary Outcome: Ingested CBD on Postprandial Metabolism Via Measurements of Insulin
Description: At the 2 randomized visits Including a Test Meal insulin Area Under the Curve was calculated from standardized intervals after ingestion of a liquid meal and a single dose of Formulation 725.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: min x mU/L
Arm/Group | Formulation 725 | Placebo
Number analyzed (Participants) | 13 | 14
min x mU/L | 7043.3 (4780.8) | 6934.75 (4556.64)

20. Primary Outcome: Ingested CBD on Postprandial Metabolism Via Measurements of Triglycerides
Description: At the 2 randomized visits Including a Test Meal triglyceride Area Under the Curve was calculated from standardized intervals after ingestion of a liquid meal and a single dose of Formulation 725.
Time Frame: as for outcome 18
Measure: Mean (Standard Deviation); unit: min x mg/dL
Arm/Group | Formulation 725 | Placebo
Number analyzed (Participants) | 10 | 14
min x mg/dL | 24978.8 (9538.7) | 30605.36 (17037.6)

21. Primary Outcome: Acute Influence of Liver Function, Alanine Aminotransferase (ALT), With the Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for alanine aminotransferase (ALT).
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: U/L
Groups:
- Placebo: Cannabidiol-free drink.
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
U/L
  0 minutes | 26.1 (10.1) | 28 (10.9) | 27.5 (8.4) | 29 (10.6) | 30.5 (11.2) | 27.7 (9.1)
  60 minutes | 26.9 (10.8) | 27.9 (10) | 29.3 (8.1) | 29.1 (9.8) | 30.4 (11) | 27.3 (8.7)
  240 minutes | 26.0 (11.2) | 28.6 (10.6) | 28.2 (7.9) | 28.7 (10.5) | 30.7 (11.5) | 27.6 (9.8)

22. Primary Outcome: Acute Influence of Liver Function, Albumin, for Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for albumin.
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
g/dL
  0 minutes | 3.6 (0.3) | 3.9 (0.3) | 3.9 (0.2) | 3.8 (0.3) | 3.8 (0.3) | 3.8 (0.3)
  60 minutes | 3.6 (0.2) | 3.8 (0.3) | 3.8 (0.3) | 3.8 (0.2) | 3.8 (0.2) | 3.8 (0.2)
  240 minutes | 3.4 (0.3) | 3.9 (0.3) | 3.9 (0.3) | 3.9 (0.2) | 4.0 (0.2) | 3.9 (0.2)

23. Primary Outcome: Acute Influence of Liver Function, Alkaline Phosphatase, With the Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for alkaline phosphatase.
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
U/L
  0 minutes | 62.1 (8.6) | 62.5 (7.9) | 63.6 (10.8) | 60.3 (6.8) | 61.9 (9.4) | 60.4 (12)
  60 minutes | 62.9 (9.8) | 60.5 (7.2) | 61.9 (11) | 61 (8.7) | 61.6 (9.3) | 60.9 (11.4)
  240 minutes | 58.8 (8.5) | 60.2 (8.0) | 61.4 (9.6) | 62.1 (9.5) | 62.3 (9.2) | 61 (12.6)

24. Primary Outcome: Acute Influence of Liver Function, Aspartate Aminotransferase, With the Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for aspartate aminotransferase.
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
U/L
  0 minutes | 28.0 (12.3) | 30.5 (4.1) | 30.2 (3.4) | 33.5 (7) | 30.6 (7.3) | 29.2 (5)
  60 minutes | 30.7 (10.4) | 30.6 (4.6) | 29.4 (8.7) | 30.9 (5.1) | 31.4 (7.4) | 28.9 (4.3)
  240 minutes | 29.4 (10.1) | 31.1 (6.8) | 30.3 (4.1) | 30.4 (5.9) | 31.9 (7.5) | 29.6 (4.4)

25. Primary Outcome: Acute Influence of Liver Function, Total Bilirubin, With the Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for total bilirubin.
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mg/dL
  0 minutes | 0.8 (0.3) | 1 (.3) | 1 (.6) | 1 (.4) | .9 (.2) | .9 (.4)
  60 minutes | 0.8 (0.3) | 0.9 (0.2) | 1 (0.6) | 1 (0.4) | 0.9 (0.2) | 0.9 (0.4)
  240 minutes | 0.8 (0.3) | 1 (0.3) | 1.1 (0.6) | 1.1 (0.4) | 1 (0.3) | 1 (0.4)

26. Primary Outcome: Acute Influence of Kidney Function, Blood Urea, With the Different Formulations of CBD.
Description: The different formulations will be standardized for CBD dose (30 mg) but will differ in their preparation (e.g. water vs. fat-soluble). At the 5 randomized Visits Not Including A Test Meal venous blood will be collected at standardized intervals and analyzed for blood urea.
Time Frame: Change from baseline at time 0, 60, 240 minutes for each formulation, visits separated by 14 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Formulation 088 | Formulation 126 | Formulation 213 | Formulation 625 | Formulation 725
Number analyzed (Participants) | 14 | 14 | 14 | 14 | 14 | 14
mg/dL
  0 minutes | 15.1 (2.7) | 14.6 (2.8) | 15.4 (4.5) | 15.4 (3.9) | 15 (3.6) | 15.9 (3.3)
  60 minutes | 14.6 (2.9) | 14.4 (2.8) | 15.1 (4.6) | 15.5 (4.1) | 14.8 (3.9) | 15.3 (3.3)
  240 minutes | 13.9 (2.5) | 13.4 (2.5) | 14 (4.2) | 14.3 (3.5) | 13.8 (3.7) | 14.1 (3.1)

27. Primary Outcome: CBD on Postprandial Metabolism Via Indirect Calorimetry
Description: At the 2 randomized visits including a Resting Metabolic Rate prior to and after ingestion of a single dose of Formulation 725 or placebo.
Time Frame: Compare 2 randomized visits Including a test meal collected during 45 minutes of resting metabolic rate
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Formulation 725 | Placebo
Number analyzed (Participants) | 14 | 14
kcal/day | 1751.7 (271.96) | 1755.31 (289.97)

ADVERSE EVENTS:
Time Frame: Throughout the seven study visits spread out over 10-12 weeks.
Groups:
- Placebo With a Meal: Separated by a minimum of 4 days.
  CBD matching Placebo: Matching Placebo
- Formulation 725 With a Meal: Separated by a minimum of 14 days.
  Cannabidiol (CBD) powder formulation: T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate (Formulation 725 water soluble. Contains sorbitol)
  Cannabidiol (CBD) Isolate in water formulation: formulation (725)
- Formulation 725 Without Meal: Separated by a minimum of 14 days.
  Cannabidiol (CBD) powder formulation: T-P-S-10 Caliper powder - 30 mg CBD in the form of 300 mg of 10% CBD isolate (Formulation 725 water soluble. Contains sorbitol)
- Formulation 088 Without a Meal: Separated by a minimum of 14 days. Cannabidiol (CBD) Oil based tincture formulation: 30 mg CBD isolate in medium-chain triglyceride (MCT) oil (1:1 ratio of CBD to Medium Chain Triglycerides oil) (Formulation 088 not water soluble)
- Formulation 126 Without a Meal: Separated by a minimum of 14 days. Cannabidiol (CBD) Gum Arabic, maltodextrin base formulation: 10% CBD Gum Arabic, maltodextrin base (Formulation 126 water soluble )
- Formulation 213 Without a Meal: Separated by a minimum of 14 days. Cannabidiol (CBD) Gum Arabic, sorbitol base formulation: 10% CBD Gum Arabic, sorbitol base (Formulation 213 water soluble)
- Formulation 625 Without a Meal: Separated by a minimum of 14 days. Pure CBD as crystalline powder (>99% purity) (Formulation 625 Not water soluble)
Arm/Group | Placebo With a Meal | Formulation 725 With a Meal | Formulation 725 Without Meal | Formulation 088 Without a Meal | Formulation 126 Without a Meal | Formulation 213 Without a Meal | Formulation 625 Without a Meal
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16

LIMITATIONS AND CAVEATS:
1. Protocol was only competed by males, even though both men and women were invited to participate in the study.
2. Commercially available meal replacements were used but are not representative of the average person's meals (i.e. solid foods).
3. A relatively small dose of CBD was administered (30mg) and does not reflect the average dose of CBD individual are self-administering. The dose is also significantly smaller than FDA approved, Epidiolex, a seizure medication.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-04-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT04971837/Prot_SAP_ICF_000.pdf